CLINICAL TRIAL: NCT03106285
Title: Effectiveness of Lactobacillus Reuteri DSM17938 Supplementation on Crying Time in Infantile Colic
Brief Title: Effectiveness of Probiotic Supplementation on Crying Time in Infantile Colic
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Cannot perform the study due to practical issues
Sponsor: BioGaia AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CSUB0130
Record Dates: First submitted 2017-03-24; First posted 2017-04-10 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Colic, Infantile
MeSH Terms: conditions — Colic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus reuteri DSM17938 (Experimental): Oil drops
  Interventions: Dietary Supplement: Lactobacillus reuteri DSM17938
- Placebo (Placebo Comparator): Oils drops
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri DSM17938 — 5 drops of active oil drops. The active dose consists of 10^8 CFU L retueri DSM17938
  Arms: Lactobacillus reuteri DSM17938
Dietary Supplement: Placebo — 5 drops of placebo drops
  Arms: Placebo

SUMMARY:
This study aims to investigate the effectiveness of Lactobacillus reuteri DSM17938 supplementation on infantile colic in Indonesian infants.

DETAILED DESCRIPTION:
Infantile colic is a problem faced by many parents and caregivers. There is no evidence that medications does help in this situation. The etiology of infantile colic is still unknown.

Lactobacillus reuteri has been shown in five studies to reduce crying time in infants diagnosed with infantile colic.

ELIGIBILITY:
Inclusion Criteria:

* otherwise healthy infants
* Infantile colic according to Roe IV criteria
* Full term infants
* Birth weight 2500 - 4000g
* Exclusively breast milk or partially breastfed
* Mothers last education degree is Senior high school

Exclusion Criteria

* Clinically suspected allergy
* Consumption of probiotics, antibiotics, PPI
* Failure to thrive

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Daily average of crying time with L reuteri vs placebo | day 7
  Daily crying diary
Daily average of crying time with L reuteri vs placebo | Day 14
  Daily crying diary
Daily average of crying time with L reuteri vs placebo | Day 21
  Daily crying diary
Daily average of crying time with L reuteri vs placebo | Day 28
  Daily crying diary

SECONDARY OUTCOMES:
Number of responder vs non-responders | baseline, day 7, 14, 21, 28
  Daily crying
Reduction of daily average crying time | baseline, day 7, 14, 21, 28
  Daily crying
Parents perception of colic severity (Diary) | baseline, day 7, 14, 21, 28
  Diary
Parents/Family quality of life (Diary) | baseline, day 7, 14, 21, 28
  Diary
Parental satisfactory (Diary) | baseline, day 7, 14, 21, 28
  Diary

CONTACTS AND LOCATIONS:
Overall Officials: Badriul Hegar, MD, PhD, Principal Investigator — RSCM, Rumah Sakit Cipto Mangunkusumo. University of Indonesia
Locations (1):
- Badriul Hegar, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No